CLINICAL TRIAL: NCT04260568
Title: How do Individuals Make Sense of and Respond to a Diagnosis of Persistent Postural Perceptual Dizziness (3PD)
Brief Title: How do Individuals Respond to a Diagnosis of 3PD
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 269319
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-02

CONDITIONS: Persistent Postural Perceptual Dizziness; Vestibular Disease; Chronic Dizziness
Keywords: PPPD; dizziness; Illness perceptions; qualitative
MeSH Terms: conditions — Vestibular Diseases; Dizziness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persistent Postural Perceptual Dizziness: Semi-structured interviews
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Patients with a diagnosis of 3PD will be sought from a multidisciplinary balance clinic. Consenting participants will take part in a face-to-face interview about their diagnosis. Data collection will consist of recorded semi-structured interviews, which will be transcribed.

SUMMARY:
No studies have explored how patients with chronic dizziness react to a diagnosis of Persistent Postural Perceptual Dizziness (3PD) and their beliefs and representations of the diagnostic label. Investigating the experience of diagnostic labelling from the perspective of patients will allow clinicians to recognise whether this is a helpful term to adopt and ways to improve the clinical consultation.

This is a qualitative study that will consist of semi-structured interviews with people with a new diagnosis of 3PD. The main objective of the study is to explore how patients react to this diagnostic label, what they understand about their diagnosis and how their own meanings affect their expectations and illness perceptions. Between 12-15 patients will be recruited from the balance clinic at Guy's Hospital, London, UK. The qualitative data will be analysed using thematic analysis which will draw on pragmatic interpretive descriptive methodology.

DETAILED DESCRIPTION:
Semi-structured interviews will be conducted with patients, following a topic guide, which may be updated iteratively during the data collection period in response to ideas that may be generated. The topic guide explores key topics: (1) the patient's narrative; (2) the illness experience; (3) receiving the diagnosis; (4) their understanding of the 3PD label and beliefs; (5) expectations of recovery and treatment; (6) psychological and emotional factors; and (7) free comments. The interviews will be audio recorded and transcribed verbatim.

Data will be analysed using inductive thematic analysis. Analysis will be conducted concurrently with data collection, allowing themes to be explored inductively as they emerge. Analysis will be performed by a multidisciplinary group consisting of a medical student, audio-vestibular physician and physiotherapist.

Analysis will be conducted with the aid of the latest version of computer software NVIVO for Windows. The medical student will lead the analysis, generating the initial codes which will then be discussed in data analysis meetings held regularly over the data collection and analysis period until the group are happy with the coding and themes generated. Data collection and analysis will be approached with critical reflexivity in order to reduce the risk of bias. The team will ensure the analysis is grounded in the data.

Patients will be included if they meet the diagnostic criteria for Persistent Postural Perceptual Dizziness (3PD). Patients will be excluded if they;

* Do not speak English or have special communication needs.
* Have cognitive impairment.
* Have acute severe psychiatric disorder (e.g. psychosis).

The investigators plan to interview a minimum of 12 participants and review the need for further interviews up to 15 participants if there are new themes developing (i.e. if the investigators have not reached data 'saturation').

ELIGIBILITY:
Inclusion Criteria:

• Patients who attend the balance clinic at Guy's Hospital and are diagnosed with Persistent Postural Perceptual Dizziness (3PD).

Exclusion Criteria:

* Patients who do not speak English or have special communication needs.
* Patients with cognitive impairment.
* Patients with acute severe psychiatric disorder (e.g. psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Persistent Postural Perceptual Dizziness (3PD)
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Experiences and views of patients with a new diagnosis of 3PD | 5 months
  To explore what people understand about the diagnosis of 3PD and how their own meanings affect their expectations and illness perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Murdin, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Louisa Murdin, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No